CLINICAL TRIAL: NCT05001191
Title: The Effect of Gentle Human Touch on Pain, Comfort and Physiological Parameters in Preterm Infants During Heel Lancing
Brief Title: The Effect of Gentle Human Touch in Preterm Infants During Heel Lancing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Yağmur Sezer Efe, Assist. Prof. Yağmur Sezer Efe, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021/453
Record Dates: First submitted 2021-07-08; First posted 2021-08-11 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Heel Lancing

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gentle Human Touch Group (Experimental)
  Interventions: Other: Gentle Human Touch
- Control group (No Intervention)

INTERVENTIONS:
Other: Gentle Human Touch — Gentle human touch, which has a pain and stress-reducing effect, is a sensitive tactile stimulus applied to the skin, without caress or massage, which provides a kind of relaxation.
  Arms: Gentle Human Touch Group

SUMMARY:
This randomized controlled experimental study is planned in order to determine the effect of gentle human touch on pain, comfort and physiological parameters in preterm infants during heel lancing matched for gestational age, gender and birth weight. The study will be performed with preterm infants hospitalized in the neonatal intensive care unit of a tertiary hospital. Ethical committee approval, institutional permission, parental written consent were obtained. The therapeutic touch will be applied 10 minutes before the heel lancing, it will continue during and after the procedure, a total of 15 minutes of sensitive touch will be applied. The practitioner will place one hand on the baby's head and the other hand on the lower abdomen covering the waist and hips of the preterm baby for 15 minutes. Before and after the study the following were evaluated in preterm infants in the gentle human touch and control group: pain, comfort and physiological parameters.

DETAILED DESCRIPTION:
This randomized controlled experimental study is planned in order to determine the effect of gentle human touch on pain, comfort and physiological parameters in preterm infants during heel lancing matched for gestational age, gender and birth weight. The research sample will consist of 50 preterm infants who meet the inclusion criteria. In the literature, the number of infants varies between 11 and 38 in different studies in which gentle human touch was applied to preterm infants. In this study, it was decided that the number of infants in the groups should be 25 according to α=95% confidence level and 90% power. In the study, it was planned to have 25 infants in the gentle human touch (GHT) and control groups. After reaching 50 preterm infants in the study, power analysis will be calculated using pain scores and it will be decided whether the sample size is sufficient or not. The infants in the GHT group will be applied gentle human touch for a total of 15 minutes, starting 10 minutes before the heel lancing and continuing during the heel lancing. The infants in the control group will not be subjected to any intervention other than their clinical routines, only observation will be made. Being 32-37 gestational age weeks, being birth weight of 1500 g and above, without a congenital anomaly, not having any disease at birth such as neonatal asphyxia, hemolytic status, metabolic disease, skin disease, patent ductus arteriosus (PDA), respiratory distress syndrome (RDS) and sepsis, no chest tube, not connected to a mechanical ventilator, not having intracranial bleeding, not taking any medication other than antibiotics and vitamin supplements, not taking opiates and sedatives within 4 hours before heel lancing, no painful intervention is applied at least one hour before the heel lancing, preterm infants whose mothers gave verbal and written consent will be included in the study. Data will be collected with the Questionnare Form, Physiological Parameters Observation Form, Neonatal Infant Pain Scale (NIPS), Premature Infant Comfort Scale (PBIC) and Pulse Oximeter.

ELIGIBILITY:
Inclusion Criteria:

* Being 32-37 gestational age weeks,
* being birth weight of 1500 g and above,
* without a congenital anomaly, not having any disease at birth such as neonatal asphyxia, hemolytic status, metabolic disease, skin disease, patent ductus arteriosus (PDA), respiratory distress syndrome (RDS) and sepsis,
* no chest tube,
* not connected to a mechanical ventilator,
* not having intracranial bleeding,
* not taking any medication other than antibiotics and vitamin supplements,
* not taking opiates and sedatives within 4 hours before heel lancing,
* no painful intervention is applied at least one hour before the heel lancing,
* preterm infants whose mothers gave verbal and written consent

Exclusion Criteria:

* having a congenital anomaly, having any disease at birth such as neonatal asphyxia, hemolytic status, metabolic disease, skin disease, patent ductus arteriosus (PDA), respiratory distress syndrome (RDS) and sepsis,
* being chest tube,
* connected to a mechanical ventilator,
* having intracranial bleeding,
* taking any medication other than antibiotics and vitamin supplements,
* taking opiates and sedatives within 4 hours before heel lancing,
* painful intervention is applied at least one hour before the heel lancing

Ages: 32 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2021-09-10 (Actual); Study Completion 2021-09-10 (Actual)

PRIMARY OUTCOMES:
Premature infants comfort scale (PICS) scores | before the heel lancing, during the heel lancing and after heel lancing 15. minute
  According to the PICS, a score between 7-35 is obtained from the scale. A high score from the scale indicates a low level of comfort. Change= (before the heel lancing, during the heel lancing and after heel lancing 15. minute )

SECONDARY OUTCOMES:
Newborn infant pain scale (NIPS) scores | before the heel lancing, during the heel lancing and after heel lancing 15. minute
  A score between 0-7 is taken from the scale. As the score increases, the severity of the pain also increases (0-2 points no pain, 3-4 points moderate pain, and >4 points severe pain). Change= (before the heel lancing, during the heel lancing and after heel lancing 15. minute )

OTHER OUTCOMES:
physiological parameters- heart rate | before the heel lancing, during the heel lancing and after heel lancing 15. minute
  heart rate. Change= (before the heel lancing, during the heel lancing and after heel lancing 15. minute )
physiological parameters- respiratory rate | before the heel lancing, during the heel lancing and after heel lancing 15. minute
  respiratory rate. Change= (before the heel lancing, during the heel lancing and after heel lancing 15. minute )
physiological parameters- oxygen saturation | before the heel lancing, during the heel lancing and after heel lancing 15. minute
  oxygen saturation. Change= (before the heel lancing, during the heel lancing and after heel lancing 15. minute )
physiological parameters- crying time | before the heel lancing, during the heel lancing and after heel lancing 15. minute
  crying time. Change= (before the heel lancing, during the heel lancing and after heel

CONTACTS AND LOCATIONS:
Overall Officials: Yağmur Sezer Efe, Assist. Prof., Principal Investigator — ErciyesUniversity
Locations (1):
- Erciyes university, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sezer Efe Y, Erdem E, Caner N, Gunes T. The effect of gentle human touch on pain, comfort and physiological parameters in preterm infants during heel lancing. Complement Ther Clin Pract. 2022 Aug;48:101622. doi: 10.1016/j.ctcp.2022.101622. Epub 2022 Jun 22. PMID 35759976